CLINICAL TRIAL: NCT01189266
Title: A Phase 1/2 Study of Suberoylanilide Hydroxamic Acid (SAHA, Vorinostat) and Local Irradiation, Followed by Maintenance SAHA in Children With Newly Diagnosed Diffuse Intrinsic Pontine Gliomas (DIPG)
Brief Title: Vorinostat and Radiation Therapy Followed by Maintenance Therapy With Vorinostat in Treating Younger Patients With Newly Diagnosed Diffuse Intrinsic Pontine Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02600; NCI-2011-02600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS0927; S12-02793; COG-ACNS0927; CDR0000683459; ACNS0927 (Other: Children's Oncology Group); ACNS0927 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH); UM1CA097452 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Diffuse Intrinsic Pontine Glioma; Gliosarcoma
MeSH Terms: conditions — Astrocytoma; Diffuse Intrinsic Pontine Glioma; Gliosarcoma | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 Phase I Vorinostat 180 mg/m^2 (Experimental): Patients in phase I received vorinostat at 180 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Vorinostat
- Arm 2 Phase 1 Vorinostat 230 mg/m^2 (Experimental): Patients received a higher dose of vorinostat at 230 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Vorinostat
- Arm 3 Phase II Evaluation Vorinostat 230 mg/m^2 (Experimental): Patients received a higher dose of vorinostat at 230 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/ day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I/II trial studies the side effects and best dose of vorinostat and to see how well it works when given together with radiation therapy followed by maintenance therapy with vorinostat in treating younger patients with newly diagnosed diffuse intrinsic pontine glioma (a brainstem tumor). Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving vorinostat together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To estimate the maximum tolerated dose (MTD) or recommend a phase 2 dose of vorinostat given concurrently with radiation in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG).

II. To define and describe the toxicities of vorinostat given concurrently with radiation in children with newly diagnosed DIPG.

III. To determine, in the context of this phase I/II trial, the anti-tumor activity of combining vorinostat with radiation, followed by maintenance vorinostat for twelve courses, in children with newly diagnosed DIPG, as measured by 12-month event-free survival (EFS) and overall survival (OS).

IV. To determine the toxicities of vorinostat for 12 additional courses after completion of vorinostat and radiation.

SECONDARY OBJECTIVES:

I. To measure non-homologous end-joining (NHEJ) activity in peripheral blood mononuclear cells (PBMCs) before treatment, at 2 weeks after starting vorinostat and radiation, and at the end of radiation.

II. To measure histone deacetylase 2 (HDAC2) levels and assess histone acetylation in PBMCs before treatment, at 2 weeks after starting vorinostat and radiation, and at the end of radiation.

III. To quantify deoxyribonucleic acid (DNA) repair proteins from the NHEJ and homologous recombination repair (HHR) pathways in tumors by either Western analysis or immunohistochemistry, if paraffin-embedded tumor is available.

OUTLINE: This is a phase I, dose-escalation study of vorinostat followed by a phase II study.

Patients receive vorinostat orally (PO) on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Patients undergo 3-dimensional (3D) conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. Patients then receive maintenance therapy comprising vorinostat PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons, are eligible without histologic confirmation; patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to be an anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, or anaplastic mixed glioma; patients with juvenile pilocytic astrocytoma, fibrillary astrocytoma, gangliogliomas, or other mixed gliomas without anaplasia are not eligible; patients with disseminated disease are not eligible, and magnetic resonance imaging (MRI) of spine must be performed if disseminated disease is suspected by the treating physician
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must not have received any prior treatment except dexamethasone and/or surgery
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 0.8 mg/dL (3 to < 6 years of age)
  * 1 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT (ALT) is 45 U/L
* Serum albumin >= 2 g/dL
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants (with the exception of valproic acid) and seizures are well controlled
* Patients must be able to swallow capsules or liquids; patients dependent on nasogastric (NG) tube feeding are not permitted to receive protocol therapy
* Enrollment must be no later than 28 days after the date of radiographic diagnosis or surgery, whichever is the later date

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients must not currently be receiving enzyme inducing anticonvulsants
* Patients on valproic acid must discontinue valproic acid for at least 2 weeks before starting protocol therapy
* Patients receiving coumadin, heparin, low-molecular weight heparin, or any other anti-coagulants are not eligible for study entry
* Patients receiving acetylsalicylic acid (ASA) (> 81 mg/day), non-steroidal anti-inflammatory drugs, clopidogrel (Plavix), dipyridamole (Persantine), or any other drug that inhibits platelet function are not eligible for study entry
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 37 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2010-08-09 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack M Su, Principal Investigator — Children's Oncology Group
Locations (180):
- United States (174):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Saint Charles Health System, Bend, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Australia (3):
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I /II study. Phase I determined Maximum Tolerated Dose between the first 2 treatment arms; zero patients completed therapy. Study was closed, then reopened to accrual. Phase II enrolled an additional 67 patients. Overall, 79 patients were enrolled but only 2 patients completed all 12 cycles of maintenance chemotherapy.
Groups:
- Arm 1, Phase I Vorinostat 180 mg/m^2: Patients in phase I received vorinostat at 180 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D conformal radiation therapy
  Intensity-Modulated Radiation Therapy: Undergo intensity-modulated radiation therapy
  Laboratory Biomarker Analysis: Correlative studies
  Vorinostat: Given PO
- Arm 2, Phase I Vorinostat 230 mg/m^2: Patients received a higher dose of vorinostat at 230 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D conformal radiation therapy
  Intensity-Modulated Radiation Therapy: Undergo intensity-modulated radiation therapy
  Laboratory Biomarker Analysis: Correlative studies
  Vorinostat: Given PO
- Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2: Patients received a higher dose of vorinostat at 230 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks). Patients underwent 3D conformal or intensity-modulated radiation therapy 5 days per week for 6 weeks. After completing concurrent vorinostat and radiation therapy, patients then received maintenance therapy comprising of vorinostat at 230 mg/m^2/ day PO on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D conformal radiation therapy
  Intensity-Modulated Radiation Therapy: Undergo intensity-modulated radiation therapy
  Laboratory Biomarker Analysis: Correlative studies
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Started | 6 | 6 | 67
Completed | 0 | 0 | 2
Not Completed | 6 | 6 | 65
Not completed — Adverse Event | 1 | 0 | 5
Not completed — Death | 0 | 0 | 5
Not completed — Lack of Efficacy | 4 | 5 | 44
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Patient refuses further therapy | 1 | 0 | 7
Not completed — No treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Phase I Vorinostat 180 mg/m^2 | Arm 2 Phase 1 Vorinostat 230 mg/m^2 | Arm 3 Phase II Evaluation Vorinostat 230 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 67 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 66 | 78
  Between 18 and 65 years | 0 | 0 | 1 | 1
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6 [4 to 16] | 9 [4 to 11] | 6 [3 to 19] | 6 [3 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 36 | 44
  Male | 2 | 2 | 31 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 15 | 16
  Not Hispanic or Latino | 5 | 5 | 51 | 61
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 8 | 8
  White | 6 | 5 | 47 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 9 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 62 | 62
  Australia | 0 | 0 | 3 | 3
  Canada | 1 | 1 | 1 | 3
  Puerto Rico | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat
Description: The dose of vorinostat in mg/sqm/day to be administered with combination chemotherapy and radiation therapy
Time Frame: Planned 7 weeks during chemoradiotherapy
Population: All patients enrolled on arm 1 and 2 who received at least 85% of the planned doses of radiation therapy and chemotherapy in the chemoradiotherapy portion of the study or who experienced DLT after after receiving at least one dose of chemoradio therapy and completing 7 weeks fo follow-up.
Measure: Number; unit: mg/m^2
Groups:
- All Phase 1 Study Participants: Arm 1, Phase 1 participants received vorinostat at 180 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks).
  Arm 2, Phase 1 participants received a higher dose of vorinostat at 230 mg/m^2/day PO on Monday through Friday weekly for the duration of radiation therapy (6-7 weeks).
Arm/Group | All Phase 1 Study Participants
Number analyzed (Participants) | 12
mg/m^2 | 230

2. Primary Outcome: Event-Free Survival
Description: Time from enrollment to disease progression, diagnosis of a second malignant neoplasm, death or last follow-up, whichever occurs first.
Time Frame: 2 years after study enrollment
Population: One patient enrolled on Arm 3 was withdrawn from study prior to the start of treatment.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 6 | 6 | 66
percent probability | 0 [0 to 0] | 0 [0 to 0] | 3.1 [0.59 to 9.6]

3. Primary Outcome: Incidence of Toxicity During Chemoradiation Therapy
Description: Proportion of patients who experience any grade 3 or higher CTC AE Version 4 adverse experience
Time Frame: Planned 7 weeks during chemoradiotherapy
Population: All patients enrolled on Arm 1 and 2 received at least one dose of chemoradiation therapy. Two patients enrolled on arm 3 did not receive protocol therapy prior to date of removal from protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 6 | 6 | 65
Participants | 5 | 2 | 24

4. Primary Outcome: Incidence of Toxicity During Maintenance Therapy
Description: Proportion of patients who experience any grade 3 or higher CTC AE Version 4 adverse experience
Time Frame: Planned 12 months of maintenance with Vorinostat
Population: All patients enrolled on arm 1 and 2 received at least one dose of maintenance therapy. Seven patients enrolled on arm 3 did not receive maintenance therapy prior to date of removal from protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 6 | 6 | 60
Participants | 6 | 4 | 39

5. Secondary Outcome: Overall Survival
Description: Time from enrollment to death or last follow-up, whichever occurs first.
Time Frame: 2 years after study enrollment
Population: One patient enrolled on Arm 3 was withdrawn from study prior to the start of treatment.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 6 | 6 | 66
percent probability | 22 [0.96 to 61] | 0 [0 to 0] | 3.1 [0.58 to 9.5]

6. Secondary Outcome: Change in H3 and H4 Acetylation Levels in PBMCs
Description: Degree of acetylation in peripheral blood monocytes will be divided into quartiles and coded as none, mild, moderation or marked.
Time Frame: Baseline to up to 7 weeks
Population: Due to budgetary issues the planned laboratory testing was not performed and no data were collected
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change in NHEJ Activity in PBMCs
Description: Descriptive statistics will be used to summarize the biological/laboratory measures and the changes in these measures across time-points.
Time Frame: Baseline to up to 7 weeks
Population: Due to budgetary issues the planned laboratory testing was not performed and no data were collected
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Levels of DNA Repair Proteins in Paraffin-embedded Blocks, Measured Via Immunohistochemistry or Western Analysis
Description: For immunohistochemistry from tumor blocks, the intensity will be graded from 1 to 3; for Western analysis, a percentage of the intensity relative to the tumor with the highest level will be measured.
Time Frame: Baseline
Population: Due to budgetary issues the planned laboratory testing was not performed and no data were collected
Arm/Group | Arm 1, Phase I Vorinostat 180 mg/m^2 | Arm 2, Phase I Vorinostat 230 mg/m^2 | Arm 3, Phase II Evaluation Vorinostat 230 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm 1 Phase I Vorinostat 180 mg/m^2 | Arm 2 Phase 1 Vorinostat 230 mg/m^2 | Arm 3 Phase II Evaluation Vorinostat 230 mg/m^2
All-Cause Mortality (participants affected / at risk) | 4/6 | 6/6 | 62/65
Serious Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 55/65
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 51/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Phase I Vorinostat 180 mg/m^2 (N=6) | Arm 2 Phase 1 Vorinostat 230 mg/m^2 (N=6) | Arm 3 Phase II Evaluation Vorinostat 230 mg/m^2 (N=65)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Death NOS (General disorders) | 3 (3) | 2 (2) | 34 (34)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 6 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 9 (10)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 9 (10)
Weight loss (Investigations) | 0 (0) | 0 (0) | 4 (4)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 11 (11) — Other, specific comments provided by the treating physician indicated all the reports were related to the patient's primary diffuse intrinsic pontine brain stem glioma.
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Phase I Vorinostat 180 mg/m^2 (N=6) | Arm 2 Phase 1 Vorinostat 230 mg/m^2 (N=6) | Arm 3 Phase II Evaluation Vorinostat 230 mg/m^2 (N=65)
Anemia (Blood and lymphatic system disorders) | 6 (10) | 6 (8) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mobitz type I (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 3 (3) | 4 (5) | 6 (6)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (6) | 5 (5)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (8) | 5 (7) | 6 (6)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (8) | 9 (10)
Fever (General disorders) | 3 (3) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 3 (3) | 5 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 2 (2)
Irritability (General disorders) | 2 (4) | 1 (1) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 2 (3) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (7) | 4 (4) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (5) | 2 (2) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 5 (5) | 2 (2) | 3 (3)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (15) | 5 (9) | 9 (9)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (8) | 4 (6) | 8 (9)
Platelet count decreased (Investigations) | 5 (10) | 5 (6) | 7 (7)
Serum amylase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Weight gain (Investigations) | 2 (2) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 2 (2) | 2 (2)
White blood cell decreased (Investigations) | 6 (12) | 4 (7) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 4 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 4 (6) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 6 (6)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 13 (13) — Other, specific comments provided by the treating physician indicated all the reports were related to the patient's primary diffuse intrinsic pontine brain stem glioma
Abducens nerve disorder (Nervous system disorders) | 2 (2) | 2 (2) | 12 (12)
Accessory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 6 (6) | 6 (6) | 19 (19)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
Dysarthria (Nervous system disorders) | 5 (6) | 1 (1) | 12 (13)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Facial nerve disorder (Nervous system disorders) | 3 (3) | 3 (3) | 12 (12)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 5 (6) | 9 (9)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 5 (6)
Hypoglossal nerve disorder (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (2) | 5 (5)
Nystagmus (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (7) | 2 (3) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT01189266/Prot_SAP_000.pdf